CLINICAL TRIAL: NCT02264236
Title: "Vaccination of Advanced-Stage Lung Cancer Patients" A Phase I/II Study of a Carbohydrate Mimotope Based Vaccine With MONTANIDETM ISA 51 VG ST Adjuvant
Brief Title: Vaccination of Advanced-Stage Lung Cancer Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inability to enroll subjects under current iteration of the protocol
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 203199; 203199 (Other: University of Arkansas for Medical Sciences)
Record Dates: First submitted 2014-10-08; First posted 2014-10-15 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- P10s-PADRE vaccine (Experimental): Subjects will be immunized by administration of either three or four doses of P10s-PADRE vaccine over a six-week period at a dose level of 500 micrograms (µg) per injection depending on the slandered of care therapy they receive for their lung cancer.
  Interventions: Biological: P10s-PADRE vaccine

INTERVENTIONS:
Biological: P10s-PADRE vaccine — P10s-PADRE vaccine combined with MONTANIDE™ ISA 51 VG "Chemotherapy" Subcutaneous injection at weeks 2, 3, 5, and 6. "3-Week Interval Immunotherapy" Subcutaneous injection at weeks 2, 3, and 4. "2-Week Interval Immunotherapy" Subcutaneous injection at weeks 3, 4, and 5.
  Other Names: Mimotope P10s-PADRE Vaccine

SUMMARY:
The overarching purpose of this study is to evaluate the clinical efficacy of an investigational agent, P10s-PADRE, a peptide mimotope-based vaccine, in combination with standard-of-care (SoC) treatment in subjects with advanced-stage (i.e., metastatic) Lung Cancer. Vaccine will consist of P10s-PADRE admixed with an adjuvant, MONTANIDETM ISA 51 VG. Up to one hundred fifty (150) subjects with advanced-stage Lung Cancer of any histologic type will be enrolled for this vaccine trial.

This single-arm, multi-site trial is designed to evaluate the therapeutic benefits of the vaccine in subjects with advanced-stage lung cancer. The primary objectives of the study are: (1) to monitor the safety and tolerability of the vaccine when it is administered in combination with SoC therapy; and (2) to determine whether immunization with vaccine can successfully elicit a robust immune response in subjects with advanced-stage lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced-stage (i.e., metastatic) Lung Cancer of any histologic type
2. (Computed Tomography) CT scans were completed within 4 weeks prior to registration
3. Age 18 years and older
4. ECOG Performance Status 0 to 2
5. White blood cell (WBC) count ≥ 3,000/mm3 within 3 weeks prior to registration
6. Platelet count ≥ 100,000/mm3 within 3 weeks prior to registration
7. Serum glutamic-pyruvic transaminase (SGPT) or alanine aminotransferase test (ALT) ≤ 2 x institutional upper limit (IUL) of normal obtained within 3 weeks prior to registration
8. Serum glutamic-oxaloacetic transaminase (SGOT) or aspartate aminotransferase test (AST) ≤ 2 x institutional upper limit (IUL) of normal obtained within 3 weeks prior to registration
9. Serum creatinine ≤ 1.8 mg/dL obtained within 3 weeks prior to registration
10. Radiation is allowed

Exclusion Criteria:

1. Active infection requiring treatment with antibiotics
2. Any other significant medical or psychiatric conditions which, in the opinion of the enrolling investigator, may interfere with consent or compliance of the treatment regimen
3. Existing diagnosis or evidence of organic brain syndrome that might preclude participation in the full protocol
4. Existing diagnosis or history of significant impairment of basal cognitive function that might preclude participation in the full protocol
5. Existing diagnosis or history of leptomeningeal disease, spinal cord compression or brain metastases unless: (a) metastases have been locally treated and have remained clinically controlled and asymptomatic for at least 14 days following treatment, AND (b) subject has no residual neurological dysfunction and has been off corticosteroids for at least 14 days prior to registration
6. Other current malignancy(s): Subjects with prior history at any time of any in situ cancer, including lobular carcinoma of the breast in situ, cervical cancer in situ, atypical melanocytic hyperplasia or Clark I melanoma in situ or basal or squamous skin cancer are eligible, provided they are disease-free at the time of registration. Subject has other malignancies have been continuously disease free for ≥ 5 years prior to the time of registration. Subjects with other malignancies are eligible if they have been continuously disease free for ≥ 5 years prior to the time of registration.
7. Active autoimmune disorders or conditions of immunosuppression; Existing autoimmune disorders or conditions of immunosuppression that have been in remission for less than 6 months.
8. Treatment with corticosteroids, including oral steroids (i.e. prednisone, dexamethasone), continuous use of topical steroid creams or ointments or any steroid-containing inhalers. Subjects who have been on systemic steroids will require a 6-week washout period. Subjects who discontinue the use of these classes of medication for at least 6 weeks prior to registration are eligible if, in the judgment of the treating physician, the subject is not likely to require these classes of drugs during the treatment period. Replacement doses of steroids for subjects with adrenal insufficiency are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with vaccine related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. | 64 weeks +/- 2 weeks per subject
  The National Cancer Institute (NCI) of the National Institutes of Health (NIH) has published standardized definitions for adverse events (AEs), known as the Common Terminology Criteria for Adverse Events (CTCAE, also called "common toxicity criteria"), to describe the severity of organ toxicity for patients receiving cancer therapy. The tables describing AEs graded in the CTCAE (version 4.0) provides a references for adverse events reporting. From grade 1 AEs being minor/low grade adverse events to grade 5 AEs being serious adverse events usually resulting in death.
Number of participants with vaccine induced immune related response. | 64 weeks +/- 2 weeks per subject

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Arnaoutakis, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States